CLINICAL TRIAL: NCT05074225
Title: Aesthetic Outcome of Electrodesiccation and Curettage vs Excision With Complex Linear Closure for Low Risk Lesions on the Trunk and Extremities: a Randomized, Blind Control Trial
Brief Title: Aesthetic Outcome of Electrodesiccation and Curettage vs Excision With Complex Linear Closure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1515118
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cutaneous Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED&C (Experimental): The ED&C arm will receive the standard ED&C care.
  Interventions: Other: Electrodesiccation and Curettage vs Excision
- Excision (Experimental): The excision arm will undergo standard excision with repair by complex linear closure.
  Interventions: Other: Electrodesiccation and Curettage vs Excision

INTERVENTIONS:
Other: Electrodesiccation and Curettage vs Excision — Factorial Assignment.
  At the follow-up visit, two blinded observers will record their scores independently using the physician observer scar assessment score instrument (POSAS).

SUMMARY:
The purpose of this study is to determine whether electrodesiccation and curettage (ED&C) versus excision with complex linear closure affects esthetic outcomes (primary outcome). As secondary outcome, we plan to look at patient quality of life measures and complications. This will be a prospective, 2-arm, randomized, evaluator-blinded clinical trial. One half of the patients will receive ED&C and the other half will receive excision with repair by complex linear closure. Three-months post-surgery, the scar will be evaluated via the patient observer scar assessment scale (POSAS), a validated scar instrument, as well as the trace-to-tape method, an objective outcome measure for linear postoperative scars. In addition, patients will be provided a validated quality of life survey to complete. Any adverse events will also be recorded.

DETAILED DESCRIPTION:
Low risk lesions on the trunk and extremities can be treated via various modalities including topical therapies, ED&C, and excision. The purpose of this study is to compare ED&C versus excision with repair by complex linear closure. The wound following ED&C will heal by second intention, meaning that there will not be any sutures placed. Complex linear closures following an excision will require two layers of sutures: a deep (subcutaneous) layer and a top (cutaneous) layer.

This study aims to investigate whether ED&C versus excision with repair by complex linear closure for low risk lesions on trunk and extremities affects cosmesis. In other words, the research team would like to determine which of the following yields a more cosmetically appealing scar: ED&C or excision with linear closure. As secondary outcomes, the research team plans to look at quality of life measures via a validated survey and complications.

There has been a prospective cohort study measuring quality of life following ED&C vs excision vs Mohs surgery1 and another prospective cohort study measuring patient reported outcomes following ED&C2. However, randomized control trials comparing the cosmesis and quality of life of these two methods appear to be lacking in current literature. The research team hopes that this study will provide new insight in cutaneous surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for treatment of low risk cutaneous neoplasms on the trunk or extremities (superficial or nodular basal cell carcinoma and squamous cell carcinoma in-situ).
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant Women
* Lesion size equal to or greater than 2 cm.
* Aggressive tumor subtypes(invasive squamous cell carcinoma (any subtype), infiltrative(sclerosing) basal cell carcinoma, micronodular basal cell carcinoma.
* Recurrent tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Scar Assessment | 3-12 months
  The primary endpoints will be (1) the score of two blinded reviewers using the patient observer scar assessment score and (2) the mean scar area to preoperative cancer area ratio using the trace-to-tape method at a three-month assessment visit.

SECONDARY OUTCOMES:
Complications | 3-12 months
  The following complications from the treatment will be evaluated: spitting sutures, dehiscence, infection, necrosis, bleeding, and hematoma.
Quality of Life Measures (DLQI) | 3-12 months
  The aim of this questionnaire is to measure how much study participant skin problem has affected their life. The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided